CLINICAL TRIAL: NCT03724487
Title: A COmmunity and Tech-Based ApproaCh for Hypertension Self-MANagement (COACHMAN)
Brief Title: A COmmunity and Tech-Based ApproaCh for Hypertension Self-MANagement
Acronym: Coachman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Carolyn Still, Assistant Professor, Frances Payne Bolton School of Nursing, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5U54MD002265-12 (NIH)
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-07

CONDITIONS: Hypertension; Self-management; Technology; Community-based Participatory Research
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coachman (Experimental): The first study condition, A COmmunity and Tech-Based ApproaCh for Hypertension Self-MANagement (COACHMAN) will be exposed to three Technology-based Interventions (TBI) accessible via smartphone and counseling from a local community nurse organization for hypertension self-management support.
  Interventions: Behavioral: Coachman
- Enhanced Usual Care (Experimental): The second study condition, Enhanced Usual Care (EUC) will be exposed to routine and standard hypertension education materials and one session on self-monitoring blood pressure.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Coachman — Coachman is comprised of: TBI and nurse counseling. TBI is comprised of: 1) web-based education modules on hypertension knowledge and skills as well as behavioral lifestyle guidance, (2) Medisafe, a smartphone medication management app to support medication adherence to antihypertensives, and (3) self-monitoring blood pressure. Participants will be exposed to nurse counseling, by registered nurses from the community, affiliated with a local nurse organization that will serve as community health workers (CHWs). The CHWs will provide informal counseling, social support, as well as follow-up phone sessions on medication adherence and monitoring blood pressure.
  Arms: Coachman
Behavioral: Enhanced Usual Care (EUC) — Standard printed education materials on hypertension management, including content on lifestyle modification and medication-taking will be provided; plus access to one web-based education (video) with information on how to self-monitoring blood pressure.
  Arms: Enhanced Usual Care

SUMMARY:
The prevalence of hypertension among U.S. adults increased from 32% to 46% and African Americans are disproportionately impacted. Self-managing hypertension presents challenges such as dealing with complex treatment regimen, including critical components of recommended hypertension treatment such as self-blood pressure monitoring, and lifestyle modifications involving diet, exercise, and tobacco cessation. African Americans with hypertension have lower adherence to self-management behavior due to multifactorial reasons. Substantial evidence has demonstrated the important role of community support in improving patients' self-management of a variety of chronic illnesses, though integrating technology in such programs are rarely offered.

The purpose of this study is to investigate the effectiveness of a community outreach program using a technology-based intervention (TBI) to support self-managing hypertension (called COACHMAN) to improve BP control.

DETAILED DESCRIPTION:
COACHMAN targets barriers to hypertension knowledge, medication adherence, problem solving skills, patient-provider communication, and social support in an effort to improve blood pressure control.

The investigators will conduct a two-arm randomized control trial (RCT) using a community participatory research approach and mixed methods to evaluate the efficacy of TBI intervention with community support (Coachman) compared to enhance usual care (ECU) among 60 African Americans with uncontrolled hypertension.

The investigators aim to:

1. Identify key content, design, and resources from a community of stakeholders, including determining facilitators and barriers of hypertension self-management among African Americans that will inform the development of COACHMAN using a mixed methods approach methods.
2. Evaluate the feasibility and acceptability of COACHMAN to improve BP control.
3. Compare the difference in BP control between Technology-based intervention (TBI) and Enhanced usual care (EUC).

ELIGIBILITY:
Inclusion Criteria:

* self-identifying as African American
* age 30 years or older
* diagnosed with hypertension, with a blood pressure >140/80 mmHg
* prescribed at least one antihypertensive medication
* able to read and understand English
* own a smartphone

Exclusion Criteria:

* history of cognitive impairment
* currently using a medication management app

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn H Still, PhD, Principal Investigator — Case Western Reserve University, School of Nursing
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: starting in Dec 2026

REFERENCES:
- [Result] Still CH, Margevicius S, Harwell C, Huang MC, Martin L, Dang PB, Wright Jnr JT. A Community and Technology-Based Approach for Hypertension Self-Management (COACHMAN) to Improve Blood Pressure Control in African Americans: Results from a Pilot Study. Patient Prefer Adherence. 2020 Nov 23;14:2301-2313. doi: 10.2147/PPA.S283086. eCollection 2020. PMID 33262580
- [Result] Still CH, Dang PB, Malaker D, Peavy TD. The Design and Rationale of a Pilot Study: A COmmunity and Tech-Based ApproaCh for Hypertension Self-MANagement (COACHMAN). J Natl Black Nurses Assoc. 2020 Jul;31(1):52-59. PMID 32853497

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coachman | Enhanced Usual Care
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Coachman: The first study condition, A COmmunity and Tech-Based ApproaCh for Hypertension Self-MANagement (COACHMAN) will be exposed to three Technology-based Interventions (TBI) accessible via smartphone and counseling from a local community nurse organization for hypertension self-management support over 12 weeks.
  TBI is comprised of: 1) web-based education modules on hypertension knowledge and skills as well as behavioral lifestyle guidance, (2) Medisafe, a smartphone medication management app to support medication adherence to antihypertensives, and (3) self-monitoring blood pressure
  Total of 30 individuals who:
  1. self-identified as African American,
  2. were 30 years of age or older,
  3. had been diagnosed with hypertension (BP >140/90 mmHg) and prescribed an antihypertensive drug,
  4. were able to read/understand English, and (5) owned a smartphone.
- Enhanced Usual Care: The second study condition, Enhanced Usual Care (EUC) will be exposed to routine and standard hypertension education materials and one session on self-monitoring blood pressure.
  Enhanced Usual Care (EUC): Standard printed education materials on hypertension management, including content on lifestyle modification and medication-taking will be provided; plus access to one web-based education (video) with information on how to self-monitoring blood pressure.
  30 individuals who:
  1. self-identified as African American,
  2. were 30 years of age or older,
  3. had been diagnosed with hypertension (BP >140/90 mmHg) and prescribed an antihypertensive drug,
  4. were able to read/understand English, and (5) owned a smartphone.
- Total: Total of all reporting groups
Arm/Group | Coachman | Enhanced Usual Care | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.97 (8.37) | 60.0 (9.49) | 59.48 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 25 | 45
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 3 | 7 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 30 | 60
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Systolic Blood pressure <130 mm Hg or diastolic Blood pressure < 80 mm Hg represents better blood pressure control.
  mm Hg
    Systolic Blood Pressure (in mmHg) | 138.51 (14.77) | 141.24 (16.92) | 139.75 (15.67)
    Diastolic Blood Pressure (in mmHg) | 81.97 (13.45) | 85.28 (12.61) | 83.72 (12.84)
PROMIS Global Health [Mean (Standard Deviation); unit: units on a scale] — Raw score range from 4-20, higher scores represent better health
  units on a scale
    PROMIS Global Health-Mental Health Subscale | 13.83 (2.83) | 13.38 (2.46) | 13.53 (2.62)
    PROMIS Global Health-Physical Health Subscale | 14.52 (2.85) | 14.28 (2.68) | 14.40 (2.79)
Education (in years) [Mean (Standard Deviation); unit: years] | 14.52 (3.38) | 14.70 (3.36) | 14.6 (3.34)
Martial Status [Count of Participants; unit: Participants]
  Single | 19 | 22 | 41
  Married | 11 | 8 | 19
Employment [Count of Participants; unit: Participants]
  Unemployed | 17 | 14 | 31
  Employed | 13 | 16 | 29
Income [Count of Participants; unit: Participants]
  <$19,999 | 8 | 8 | 16
  $20,000 - $59,999 | 9 | 11 | 20
  >$60,000 | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Blood Pressure
Description: The primary outcome was a change (reduction) in both the systolic and diastolic blood pressure from baseline to 12 weeks, in which the 12 weeks mean systolic minus the baseline systolic were calculated. The same for 12 week diastolic BP minus the baseline diastolic BP were calculated for a mean change score. The change score (number) can range from no change (0) to a 10 point reduction in blood pressure.
Time Frame: baseline and 12 weeks
Population: Per protocol population, completing 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Coachman: This group was exposed to three Technology-based Interventions (TBI) accessible via smartphone and counseling from a local community nurse organization for hypertension self-management support.
Arm/Group | Coachman | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 30 | 30
mm Hg
  Systolic Blood Pressure Change from baseline at 12 weeks | 0.55 (1.84) | -2.17 (0.51)
  Diastolic Blood Pressure Change from baseline at 12 weeks | -0.80 (2.00) | -1.04 (0.55)

2. Primary Outcome: Change in PROMIS Global Health-10 [Health-related Quality of Life]
Description: Change in PROMIS Global Health-10 score (two subscales- Mental and Physical Health) from baseline to 12 weeks. Raw scores range from 4-20, higher scores represent better health. The change score is calculated as a mean difference between the two scores: at baseline and at 12 weeks. Scores are reported as a change value number, on a continuous number scale, that can be negative or positive (0 to 1, higher number better health).
Time Frame: Baseline and 12-weeks
Population: Per protocol population, completing the baseline and 12-month visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Coachman | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 30 | 30
score on a scale
  Chang in PROMIS Global Health-Metal Health Subscale | 0 (0.30) | 0.34 (0.93)
  Changes in PROMIS Global Health-Physical Health Subscale | -0.11 (0.16) | -0.11 (0.09)

3. Secondary Outcome: Achieved Blood Pressure Target of < 130/80 mm Hg at 12 Weeks
Description: Achieved Blood Pressure target is defined as the rate of participants that have a blood pressure of at the end of 12 weeks, < 130 mm Hg for systolic blood pressure and <80 mmHg diastolic blood pressure, in the intervention group. Percentage of individuals that achieved blood pressure target can range from 0 -100%
Time Frame: 12 weeks
Population: Per protocol population, individuals in the Intervention Group
Measure: Number; unit: percentage of particioants
Arm/Group | Coachman
Number analyzed (Participants) | 30
percentage of particioants | 22

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Coachman | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coachman (N=30) | Enhanced Usual Care (N=30)
Hypertensive Crisis or urgency (Vascular disorders) | 0 (0) | 0 (0) — blood pressure readings that are 180/110 mm Hg or higher -

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT03724487/Prot_SAP_000.pdf